CLINICAL TRIAL: NCT03845140
Title: An Open Label, Phase III Efficacy and Safety Study of L-PZQ ODT in Schistosoma Infected Children 3 Months to 6 Years of Age, Including a 2:1 Randomized, Controlled Cohort of Schistosoma Mansoni Infected Children 4 to 6 Years of Age Treated With L PZQ ODT or Commercial PZQ (Biltricide®)
Brief Title: L-PZQ ODT in Schistosoma Infected Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS200661_0003
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-09

CONDITIONS: Schistosomiasis
Keywords: Schistosomiasis; Children; L-praziquantel; Biltricide®
MeSH Terms: conditions — Schistosomiasis | interventions — Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1a: 4 to 6 years L-PZQ ODT 50 mg/kg (Experimental): Participants aged 4 to 6 years infected with Schistosoma (S.) mansoni received Levorotatory enantiomer of praziquantel (L-PZQ) orodispersible tablets (ODT) (150 milligrams [mg]) orally at a dose of 50 milligram per kilogram (mg/Kg) as a single oral dose after food-intake on Day 1.
  Interventions: Drug: L-PZQ ODT 50 mg/kg
- Cohort 1b: 4 to 6 years Biltricide® 40 mg/kg (Active Comparator): Participants aged 4 to 6 years infected with S. mansoni received Racemate Praziquantel tablets (Biltricide®) (600 mg) orally at a dose of 40 mg/kg as a single oral dose after food-intake on Day 1.
  Interventions: Drug: Biltricide®
- Cohort 2: 2 to 3 years L-PZQ ODT 50 mg/kg (Experimental): Participants aged 2 to 3 years infected with S. mansoni received L-PZQ ODT (150 mg) tablet orally at a dose of 50 mg/kg as a single oral dose after food-intake on Day 1.
  Interventions: Drug: L-PZQ ODT 50 mg/kg
- Cohort 3: 3 to 24 months L-PZQ ODT 50 mg/kg (Experimental): Participants aged 3 to 24 months infected with S. mansoni received L-PZQ ODT (150 mg) tablet orally at a dose of 50 mg/kg as a single oral dose after food-intake on Day 1.
  Interventions: Drug: L-PZQ ODT 50 mg/kg
- Cohort 4a: 3 months to 6 years L-PZQ ODT 50 mg/kg (Experimental): Participants aged 3 months to 6 years infected with S. haematobium received L-PZQ ODT (150 mg) tablet orally at a dose of 50 mg/kg as a single oral dose after food-intake on Day 1.
  Interventions: Drug: L-PZQ ODT 50 mg/kg
- Cohort 4b: 3 months to 6 years L-PZQ ODT 60 mg/kg (Experimental): Participants aged 3 months to 6 years infected with S. haematobium received L-PZQ ODT (150 mg) tablet orally at a dose of 60 mg/kg as a single oral dose after food-intake on Day 1.
  Interventions: Drug: L-PZQ ODT 60 mg/kg

INTERVENTIONS:
Drug: L-PZQ ODT 50 mg/kg — Participants received single oral dose of L-PZQ ODT 50 mg/Kg on Day 1.
  Arms: Cohort 1a: 4 to 6 years L-PZQ ODT 50 mg/kg; Cohort 2: 2 to 3 years L-PZQ ODT 50 mg/kg; Cohort 3: 3 to 24 months L-PZQ ODT 50 mg/kg; Cohort 4a: 3 months to 6 years L-PZQ ODT 50 mg/kg
Drug: Biltricide® — Participants received single oral dose of Biltricide® 40 mg/kg on Day 1.
  Arms: Cohort 1b: 4 to 6 years Biltricide® 40 mg/kg
Drug: L-PZQ ODT 60 mg/kg — Participant received single oral dose of L-PZQ ODT 60 mg/kg on Day 1.
  Arms: Cohort 4b: 3 months to 6 years L-PZQ ODT 60 mg/kg

SUMMARY:
The study would evaluate the safety and efficacy of L-praziquantel orodispersible (L-PZQ ODT) tablets in Schistosoma infected children aged 3 months to 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Age of the participant is 4 to 6 years of age (Cohorts 1 and 4), 2 to 3 years of age (Cohorts 2 and 4) 3 to less than 24 months of age (Cohorts 3 and 4)
* Participants are; Schistosoma (S.) mansoni positive (Cohorts 1, 2, and 3); diagnosis defined as positive egg counts in stool greater than or equal to ( >=) 1 egg per 1 occasion) according to World Health Organization (WHO) classification [1]: light (1 to 99 eggs per gram of feces), moderate (100 to 399 eggs per gram of feces) and heavy (>= 400 eggs per gram of feces) infections; S. haematobium positive (Cohort 4); diagnosis defined as positive egg counts in urine (>= 1 egg per 10 milliliter(mL) urine) according to WHO classification (Prevention and Control of Schistosomiasis and Soil Transmitted Helminthiasis. WHO Technical Report Series No. 912. WHO, Geneva, Switzerland, 2002).light (less than (<) 50 eggs per 10 mL of urine) and heavy (>=50 eggs per 10 mL of urine) infections
* Participants have a minimum body weight of 8.0 Kilograms (Kg) in 2 to 6 years of age children and 5.0 Kg in 3 months to < 24 months of age infants and toddlers
* Parent's or guardian/legally authorized representative's ability to communicate well with the Investigator and his/her delegate, to understand the protocol requirements and restrictions, and to be willing to have their children comply with the requirements of the entire study, that is:

  * To be examined by a study physician at screening and 17 to 21 days after treatment
  * To provide stool samples at screening and 17 to 21 days after treatment
  * To provide urine samples at screening and 17 to 21 days after treatment
  * To provide venous blood samples for laboratory assessments
  * To be housed in the clinic for 12 to 24 hours
  * To provide venous blood samples for pharmacokinetics (PK) assessments (for participants in the PK subset)
* Participants have a minimum hemoglobin level of 10 gram per deciliter

Exclusion Criteria:

* Participants with following medical conditions are excluded from the study; Findings in the clinical examination and/or laboratory safety examination on the treatment day, that in the opinion of the Investigator constitute a risk or a contraindication for the child's participation in the study or that could interfere with the study objectives, conduct or evaluation. This includes but is not restricted to bacterial or viral infections, such as dysentery, gastroenteritis, ascites, jaundice, etc.; Participants with seizures and/or medical history of seizures and/or other signs of potential central nervous system involvement; Participants with known cysticercosis, or with signs or symptoms (for example: subcutaneous nodules) suggestive of cysticercosis; Participants with an acute infection or other acute illness within the 7 days prior to study screening; Debilitating illness such as tuberculosis, malnutrition, etc.
* Treatment with PZQ within the 4 weeks prior to the study screening
* Concomitant treatment (within 2 weeks prior to enrollment) with medication that might affect the metabolism of PZQ, such as certain anti epileptics (for example: carbamazepine or phenytoin), glucocorticosteroids (for example: dexamethasone), chloroquine, rifampicin or cimetidine (see Biltricide® Summary of Product Characteristics [SmPC])
* Treatment within the 2 weeks prior to the study screening with anti malarial medications
* For infants and toddlers being breast fed, treatment of the mothers/wet nurses with PZQ in the 3 days prior to PZQ ODT administration
* Participation in any clinical study within 4 weeks prior to administration of PZQ ODT, or anticipated at any time until completion of the End of study visit
* Participants with marked increases of the liver enzymes: alanine aminotransferase and/or aspartate aminotransferase above 3 times the upper limit of normal (ULN); total bilirubin level above 1.5 times the ULN
* Participants with hepatosplenic schistosomiasis
* Fever, defined as temperature above 37.5 degree Celsius axillary or oral mixed S. haematobium and S. mansoni infections

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 288 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (2):
- Universitè de Cocody, Abidjan, Côte d’Ivoire
- Kemri Kisumu, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Derived] N'Goran EK, Odiere MR, Assande Aka R, Ouattara M, Aka NAD, Ogutu B, Rawago F, Bagchus WM, Bodding M, Kourany-Lefoll E, Tappert A, Yin X, Bezuidenhout D, Badenhorst H, Huber E, Dalken B, Haj-Ali Saflo O. Efficacy, safety, and palatability of arpraziquantel (L-praziquantel) orodispersible tablets in children aged 3 months to 6 years infected with Schistosoma in Cote d'Ivoire and Kenya: an open-label, partly randomised, phase 3 trial. Lancet Infect Dis. 2023 Jul;23(7):867-876. doi: 10.1016/S1473-3099(23)00048-8. Epub 2023 Mar 6. PMID 36893784
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200661_0003
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Started | 100 | 50 | 30 | 18 | 30 | 60
Completed | 100 | 49 | 30 | 18 | 30 | 60
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Participant travelled outside study area | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population (SAF) included all participants who received 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg | Total
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.4 (0.69) | 5.5 (0.83) | 3.0 (0.59) | 1.4 (0.43) | 4.6 (1.49) | 5.1 (1.51) | 4.8 (1.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 21 | 16 | 11 | 9 | 28 | 137
  Male | 48 | 29 | 14 | 7 | 21 | 32 | 151
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 100 | 50 | 30 | 18 | 30 | 60 | 288
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1a and Cohort 1b: Number of Participants With Clinical Cure Determined by Kato-Katz Method
Description: Clinical cure was defined as no parasite egg in the stool at Week 3 as determined by the Kato-Katz method. Number of participants with clinical cure were reported.
Time Frame: at Week 3
Population: Modified intent to treat analysis population (mITT) included all enrolled participants who received one dose of treatment and had baseline measurement, excluding those who used anti-malaria treatment after enrollment. Only 1 participant from Cohort 1b was lost to follow-up and was imputed as non-cured.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg
Number analyzed (Participants) | 98 | 48
Participants | 86 | 39

2. Secondary Outcome: Cohort 2 and Cohort 3: Number of Participants With Clinical Cure Determined by Kato-Katz Method
Description: as for outcome 1
Time Frame: at Week 3
Population: mITT included all enrolled participants who received one dose of treatment and had baseline measurement, excluding those who used anti-malaria treatment after enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg
Number analyzed (Participants) | 29 | 18
Participants | 27 | 17

3. Secondary Outcome: Cohort 4a and Cohort 4b: Number of Participants With Clinical Cure Determined by Urine Filtration Technique
Description: Clinical cure was defined as no parasite egg in the urine samples at follow up as determined by the urine filtration technique. Number of participants with clinical cure were reported.
Time Frame: Week 3 and Week 5
Population: mITT included all enrolled participants who received one dose of treatment and had baseline measurement, excluding those who used anti-malaria treatment after enrollment. Here "Number Analyzed" signifies those participants who were evaluated at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 29 | 58
Participants
  Week 3 | 17 | 50
  Week 5: number analyzed (Participants) | 0 | 58
  Week 5 |  | 55

4. Secondary Outcome: Cohort 1a, Cohort 1b, Cohort 2 and Cohort 3: Egg Reduction Rate (Percent [%]) Determined by Kato-Katz Method
Description: Percentage of reduction in group mean egg count was calculated as relative difference between the post-treatment arithmetic mean egg count and pre-treatment arithmetic mean egg count at baseline count, (pre-treatment mean egg count minus post-treatment mean egg count divided by pre-treatment mean egg count) *100. Egg counts were determined by the Kato-Katz method.
Time Frame: Pre-treatment, Week 3 post-treatment
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percent reduction in egg count
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg
Number analyzed (Participants) | 98 | 48 | 29 | 18
percent reduction in egg count | 99.5 [98.8 to 99.9] | 99.2 [97.6 to 99.8] | 88.5 [56.4 to 100.0] | 95.6 [77.0 to 100.0]

5. Secondary Outcome: Cohort 4a and Cohort 4b: Egg Reduction Rate (Percent [%]) Determined by Urine Filtration Technique
Description: Percentage of reduction in group mean egg count was calculated as relative difference between the post-treatment arithmetic mean egg count and pre-treatment arithmetic mean egg count at baseline count, (pre-treatment mean egg count minus post-treatment mean egg count divided by pre-treatment mean egg count) *100. Egg counts were determined by the urine filtration technique.
Time Frame: Pre-treatment, Weeks 3 and 5 post-treatment
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percent reduction in egg count
Arm/Group | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 29 | 58
percent reduction in egg count
  Week 3 | 99.4 [98.8 to 99.8] | 99.2 [98.2 to 99.8]
  Week 5: number analyzed (Participants) | 0 | 58
  Week 5 |  | 99.3 [97.6 to 100.0]

6. Secondary Outcome: Cohort 1a, Cohort 1b, Cohort 2, and Cohort 3: Number of Participants With Clinical Cure Determined by Point-of-Care Circulating Cathodic Antigen (POC-CCA) Test
Description: Clinical cure is defined as absence of test line in the POC-CCA test cassette (that is no Schistosoma antigens detected). Number of participants with clinical cure were reported.
Time Frame: at Week 3
Population: mITT analysis population included all enrolled participants who received one dose of treatment and had baseline measurement, excluding those who used anti-malaria treatment after enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg
Number analyzed (Participants) | 98 | 48 | 29 | 18
Participants | 63 | 26 | 18 | 13

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs and Treatment-Related TEAEs
Description: Adverse Event (AE) was defined any untoward medical occurrence in a participant administered with a study drug, which does not necessarily had a causal relationship with this treatment. Serious AE was defined AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect. TEAEs: TEAEs were defined as those events with onset dates/time occurring after study intervention administration or events that worsen after study intervention administration. TEAEs included serious TEAEs and non-serious TEAEs. Treatment-related TEAEs: reasonably related to the study intervention.
Time Frame: up to Day 40
Population: SAF anlysis population included all participants who received 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
Participants
  Participants with TEAEs | 66 | 31 | 20 | 14 | 9 | 28
  Participants with serious TEAEs | 0 | 0 | 0 | 0 | 0 | 1
  Participants with treatment-related TEAEs | 31 | 14 | 16 | 4 | 0 | 5

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) by Severity According to Qualitative Toxicity Scale
Description: Severity of TEAEs were graded using Qualitative Toxicity Scale, as follows: Mild: Participant is aware of the event or symptom, but the event or symptom is easily tolerated; Moderate: Participant experiences sufficient discomfort to interfere with or reduce his or her usual level of activity; Severe: Significant impairment of functioning: the participant is unable to carry out his or her usual activities. Number of participants with TEAEs by severity were reported.
Time Frame: up to Day 40
Population: SAF anlysis population included all participants who received 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
Participants
  Mild | 57 | 27 | 19 | 14 | 5 | 21
  Moderate | 21 | 8 | 9 | 2 | 4 | 12
  Severe | 1 | 1 | 1 | 0 | 0 | 1

9. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameter: erythrocytes mean corpuscular hemoglobin. Change from baseline in hematology parameter: erythrocytes mean corpuscular hemoglobin at Day 1 were reported.
Time Frame: Baseline, Day 1
Population: SAF included all participants who received 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: picogram
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
picogram | -0.12 (1.273) | 0.20 (0.665) | 0.18 (0.348) | 0.34 (0.699) | 0.02 (0.325) | 0.30 (1.046)

10. Secondary Outcome: Change From Baseline in Hematology Parameters: Erythrocytes Mean Corpuscular Hemoglobin (HGB) Concentration and Hemoglobin
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameters: erythrocytes mean corpuscular HGB concentration and hemoglobin. Change from baseline in hematology parameters: erythrocytes mean corpuscular HGB concentration and hemoglobin at Day 1 were reported.
Time Frame: Baseline, Day 1
Population: SAF included all participants who received 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
gram per liter (g/L)
  Erythrocytes Mean Corpuscular HGB Concentration | -0.6 (10.95) | 3.1 (9.97) | 5.2 (13.85) | 3.9 (11.25) | 4.5 (6.52) | 1.0 (11.82)
  Hemoglobin | -0.8 (8.26) | -0.0 (11.56) | -4.4 (10.29) | 1.1 (7.22) | -0.1 (6.89) | 0.8 (7.43)

11. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameter: erythrocytes mean corpuscular volume. Change from baseline in hematology parameter: erythrocytes mean corpuscular volume at Day 1 were reported.
Time Frame: Baseline, Day 1
Population: SAF included all participants who received 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
femtoliters | -0.24 (2.657) | -0.04 (1.247) | -0.06 (0.905) | 0.16 (2.101) | -0.88 (0.948) | 0.61 (1.381)

12. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameter: erythrocytes. Change from baseline in hematology parameter: erythrocytes at Day 1 were reported.
Time Frame: Baseline, Day 1
Population: SAF included all participants who received 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
10^12 cells per liter | -0.003 (0.3245) | -0.061 (0.3792) | -0.240 (0.5650) | -0.044 (0.3724) | 0.001 (0.2921) | -0.028 (0.4000)

13. Secondary Outcome: Change From Baseline in Hematology Parameters: Hematocrit, Lymphocytes/Leukocytes, Mixed Cells/Leukocytes, Neutrophils/Leukocytes
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameters: hematocrit, lymphocytes/leukocytes, mixed cells/leukocytes, neutrophils/leukocytes. Change from baseline in hematology parameters: hematocrit, lymphocytes/leukocytes, mixed cells/leukocytes, neutrophils/leukocytes at Day 1 were reported.
Time Frame: Baseline, Day 1
Population: SAF included all participants who received 1 dose of study treatment. Here "Number Analyzed" signifies those participants who were evaluated in specified categories.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
percentage of cells
  Hematocrit | 0.075 (3.3856) | -0.434 (3.0010) | -1.787 (3.9566) | -0.144 (2.6203) | -0.400 (2.3799) | 0.103 (3.0415)
  Lymphocytes/Leukocytes | 4.35 (10.617) | 1.69 (9.171) | 0.44 (10.390) | 6.13 (7.579) | 3.75 (7.973) | 5.82 (8.456)
  Mixed Cells/Leukocytes | -1.35 (6.526) | 0.45 (7.579) | 0.07 (4.816) | 0.19 (4.597) | 1.87 (4.278) | -1.19 (6.436)
  Neutrophils/Leukocytes: number analyzed (Participants) | 90 | 46 | 26 | 18 | 6 | 60
  Neutrophils/Leukocytes | -2.01 (13.738) | -3.03 (13.733) | 0.15 (13.430) | -6.32 (8.848) | -11.68 (8.228) | -4.60 (11.336)

14. Secondary Outcome: Change From Baseline in Hematology Parameters: Leukocytes and Platelets
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the hematology parameters: leukocytes and platelets. Change from baseline in hematology parameters: leukocytes and platelets at Day 1 were reported.
Time Frame: Baseline, Day 1
Population: SAF included all participants who received 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
10^9 cells per liter
  Leukocytes | -0.357 (2.2500) | -0.512 (2.3055) | -0.967 (1.9043) | 0.317 (2.1385) | -0.390 (1.9805) | 0.340 (1.9324)
  Platelets | -21.2 (56.04) | -24.5 (39.08) | -28.6 (61.75) | 49.7 (170.67) | -10.0 (33.12) | -14.0 (62.78)

15. Secondary Outcome: Change From Baseline in Chemistry Parameters: Alanine Aminotransferase and Aspartate Aminotransferase
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the chemistry parameters: Alanine Aminotransferase and Aspartate Aminotransferase. Change from baseline in chemistry parameters: Alanine Aminotransferase and Aspartate Aminotransferase at Day 1 were reported.
Time Frame: Baseline, Day 1
Population: SAF included all participants who received 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
units per liter (U/L)
  Alanine Aminotransferase | -1.91 (5.447) | -1.23 (6.245) | -2.03 (3.945) | -0.40 (5.959) | -1.27 (2.532) | -1.57 (3.614)
  Aspartate Aminotransferase | -2.50 (9.271) | -0.59 (12.759) | -2.55 (8.910) | 4.41 (27.941) | -2.87 (4.805) | -1.93 (4.430)

16. Secondary Outcome: Change From Baseline in Chemistry Parameters: Bilirubin, Creatinine and Direct Bilirubin
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the chemistry parameters: bilirubin, creatinine and direct bilirubin. Change from baseline in chemistry parameters: bilirubin, creatinine and direct bilirubin at Day 1 were reported.
Time Frame: Baseline, Day 1
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: micromole per liter (mcmol/L)
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
micromole per liter (mcmol/L)
  Bilirubin: number analyzed (Participants) | 56 | 27 | 6 | 6 | 0 | 0
  Bilirubin | -1.48 (3.056) | -0.22 (2.531) | 0.25 (3.651) | -1.62 (3.075) |  |
  Creatinine | 4.565 (10.7273) | 6.386 (13.9391) | 3.340 (16.7903) | 1.644 (8.2799) | 9.733 (10.7220) | 6.967 (13.1561)
  Direct Bilirubin: number analyzed (Participants) | 44 | 23 | 24 | 12 | 30 | 60
  Direct Bilirubin | 0.09 (0.937) | 0.06 (0.278) | 0.05 (0.219) | -0.04 (0.144) | -0.05 (0.523) | 0.07 (0.453)

17. Secondary Outcome: Change From Baseline in Chemistry Parameter: C Reactive Protein
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the chemistry parameter: C reactive protein. Change from baseline in chemistry parameter: C reactive protein at Day 1 were reported.
Time Frame: Baseline, Day 1
Population: SAF included all participants who received 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
milligram per liter (mg/L) | 0.411 (9.6546) | 0.004 (3.5448) | -0.336 (3.8792) | 0.872 (4.6025) | -0.588 (4.2572) | 0.283 (3.3653)

18. Secondary Outcome: Change From Baseline in Chemistry Parameters: Glucose, Urea and Urea Nitrogen
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the chemistry parameters: glucose, urea and urea nitrogen. Change from baseline in chemistry parameters: glucose, urea and urea nitrogen at Day 1 were reported.
Time Frame: Baseline, Day 1
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
millimole per liter (mmol/L)
  Glucose | -0.056 (1.2426) | 0.277 (1.3265) | 0.207 (1.2011) | -0.354 (1.4042) | -0.070 (1.0867) | -0.052 (1.4386)
  Urea: number analyzed (Participants) | 56 | 27 | 6 | 6 | 0 | 0
  Urea | 0.061 (0.1159) | 0.087 (0.0691) | 0.082 (0.0611) | 0.043 (0.0528) |  |
  Urea Nitrogen: number analyzed (Participants) | 44 | 23 | 24 | 12 | 30 | 60
  Urea Nitrogen | 1.443 (1.2279) | 1.257 (1.1638) | 2.017 (1.7597) | 0.614 (0.9841) | 1.966 (1.2305) | 2.432 (1.3376)

19. Secondary Outcome: Change From Baseline in Chemistry Parameter: Total Protein
Description: Blood samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the chemistry parameter: total Protein. Change from baseline in chemistry parameter: total Protein at Day 1 were reported.
Time Frame: Baseline, Day 1
Population: SAF included all participants who received 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: gram per liter (g/L)
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
gram per liter (g/L) | -5.20 (5.001) | -6.32 (5.018) | -6.22 (7.241) | 0.16 (4.918) | -3.40 (5.308) | -3.18 (4.959)

20. Secondary Outcome: Change From Baseline in Urinalyses Parameter: Specific Gravity of Urine
Description: Urine samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the urinalyses parameters: specific gravity. Change from baseline in urinalyses parameter: specific gravity Day 1 was reported.
Time Frame: Baseline, Day 1
Population: SAF included all participants who received 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
ratio | 0.0066 (0.00797) | 0.0064 (0.00722) | 0.0060 (0.00781) | 0.0039 (0.00932) | 0.0047 (0.00787) | 0.0091 (0.00704)

21. Secondary Outcome: Change From Baseline in Urinalyses Parameter: Potential of Hydrogen (pH) of Urine
Description: Urine samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the urinalyses parameter: pH. Change from baseline in urinalyses parameter: pH at Day 1 was reported.
Time Frame: Baseline, Day 1
Population: SAF included all participants who received 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
pH | -0.33 (1.176) | -0.54 (1.068) | -0.50 (1.017) | -0.11 (0.654) | -0.42 (0.872) | -0.43 (0.899)

22. Secondary Outcome: Change From Baseline in Urinalyses Parameter: Urobilinogen
Description: Urine samples were collected in a fasted condition (after a fast of at least 12 hours) to analyze the urinalyses parameter: urobilinogen. Change from baseline in urinalyses parameter: urobilinogen at Day 1 were reported.
Time Frame: Baseline, Day 1
Population: SAF included all participants who received 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
mcmol/L | 0.01 (4.069) | 0.19 (4.387) | 0.48 (2.355) | 0.00 (0.000) | -0.03 (0.146) | 0.01 (0.090)

23. Secondary Outcome: Change From Baseline in Vital Signs: Diastolic Blood Pressure and Systolic Blood Pressure
Description: Diastolic blood pressure and systolic blood pressure were measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Change from baseline in vital signs: diastolic blood pressure and systolic blood pressure at Week 3 were reported.
Time Frame: Baseline, Week 3
Population: SAF included all participants who received 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
millimeters of mercury (mmHg)
  Diastolic Blood Pressure | 2.7 (10.92) | 2.0 (9.49) | 2.9 (10.58) | -1.3 (10.27) | 1.2 (12.49) | 4.1 (11.73)
  Systolic Blood Pressure | -0.5 (12.37) | -1.4 (12.17) | 0.3 (12.58) | 0.8 (8.06) | -1.8 (9.78) | 3.7 (12.07)

24. Secondary Outcome: Change From Baseline in Vital Signs: Pulse Rate
Description: Pulse rate was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Change from baseline in vital sign: pulse rate at Week 3 was reported.
Time Frame: Baseline, Week 3
Population: SAF included all participants who received 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
beats per minute | -1.8 (14.65) | -2.6 (11.90) | -4.1 (20.46) | -9.6 (20.74) | -3.7 (18.78) | -1.7 (11.90)

25. Secondary Outcome: Change From Baseline in Vital Sign: Respiratory Rate
Description: Respiratory rate was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Change from baseline in vital sign: respiratory rate at Week 3 was reported.
Time Frame: Baseline, Week 3
Population: SAF included all participants who received 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
breaths per minute | 0.5 (4.09) | -0.1 (3.63) | -1.0 (2.98) | -3.4 (8.91) | -2.6 (3.85) | -0.9 (4.02)

26. Secondary Outcome: Change From Baseline in Vital Signs: Temperature
Description: Temperature was measured after at least 5 minutes of rest for the participant in a quiet sitting without distractions. Change from baseline in vital sign: temperature at Week 3 was reported.
Time Frame: Baseline, Week 3
Population: SAF included all participants who received 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
degree Celsius | -0.02 (0.482) | -0.04 (0.529) | 0.21 (0.734) | -0.10 (0.484) | -0.01 (0.529) | 0.08 (0.427)

27. Secondary Outcome: Number of Participants With Reaction to Study Intervention Administration
Description: Reaction to study intervention administration were recorded to describe tolerability as assessed by nurse/site staff for all children enrolled in the study. Reactions categorized as spitting, crying, diarrheas, sleepiness, abdominal pain, fever, vomiting and other. Number of participants with reaction to study intervention administration reported.
Time Frame: Day 1
Population: SAF anlysis population included all participants who received 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 100 | 50 | 30 | 18 | 30 | 60
Participants
  Crying | 1 | 4 | 8 | 8 | 2 | 2
  Spitting | 1 | 3 | 6 | 6 | 0 | 3
  Diarrhoea | 16 | 3 | 4 | 2 | 0 | 2
  Sleepiness | 7 | 3 | 7 | 2 | 0 | 1
  Abdominal pain | 21 | 9 | 9 | 0 | 0 | 2
  Fever | 1 | 1 | 0 | 0 | 0 | 0
  Vomiting | 7 | 4 | 4 | 1 | 0 | 0
  Other | 3 | 1 | 0 | 0 | 0 | 1

28. Secondary Outcome: Cohort 1a, Cohort 1b, Cohort 4a and Cohort 4b: Palatability Assessment Based on Visual Analog Scale (VAS) Score
Description: Palatability of the study intervention was assessed using a human gustatory sensation test (100-millimeter [mm] visual analog scale [VAS]) incorporating a facial hedonic scale, where lower score (0) indicates "not acceptable/not liked at all" and higher score (100) indicates "very acceptable/liked very much".
Time Frame: Day 1
Population: SAF included all participants who received 1 dose of study treatment. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 73 | 34 | 13 | 35
score on a scale | 84.0 [54.0 to 91.0] | 50.0 [26.0 to 87.0] | 88.0 [69.0 to 91.0] | 88.0 [79.0 to 92.0]

29. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Praziquantel (PZQ) Enantiomers: R-PZQ and S-PZQ
Description: Cmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours post-dose
Population: The Pharmacokinetic Analysis Population (PKP) is a subset of the SAF population and consisted of all participants who received at least one dose of active Investigational Medicinal Product (IMP) and provide at least one measurable post-dose concentration.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 17 | 10 | 9 | 2 | 14 | 15
nanogram per milliliter (ng/mL)
  R-PZO | 347 (281.4) | 59.3 (60.39) | 1470 (1326) | NA (NA) — Mean and standard deviation was not calculated for participants fewer than 3 as per planned analysis. | 523 (667.7) | 300 (239.7)
  S-PZO | 1.27 (2.834) | 343 (298.9) | 0.00 (0.000) | NA (NA) — Mean and standard deviation was not calculated for participants fewer than 3 as per planned analysis. | 0.00 (0.000) | 0.360 (1.394)

30. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Praziquantel (PZQ) Enantiomers: R-PZQ and S-PZQ
Description: Tmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours post-dose
Population: PKP analysis population is a subset of the SAF population and consisted of all participants who received at least one dose of active IMP and provide at least one measurable post-dose concentration.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 17 | 10 | 9 | 2 | 14 | 15
hours
  R-PZO | 02.00 [0.500 to 8.00] | 01.00 [0.00 to 12.0] | 03.00 [01.00 to 12.0] | NA [NA to NA] — Median and Full range was not calculated for participants fewer than 3 as per planned analysis. | 1.50 [0.500 to 6.02] | 03.00 [0.500 to 8.02]
  S-PZO | 0.00 [0.00 to 4.00] | 2.49 [0.500 to 12.0] | 0.00 [0.00 to 8.00] | NA [NA to NA] — Median and Full range was not calculated for participants fewer than 3 as per planned analysis. | 0.00 [0.00 to 5.00] | 0.00 [0.00 to 5.00]

31. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Praziquantel (PZQ) Enantiomers: R-PZQ and S-PZQ
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours post-dose
Population: PKP analysis population is a subset of the SAF population and consisted of all participants who received at least one dose of active IMP and provide at least one measurable post-dose concentration. Here "Number Analyzed" signifies those participants who were evaluated in specified categories.
Measure: Mean (Standard Deviation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
Number analyzed (Participants) | 17 | 10 | 9 | 2 | 14 | 15
hours*nanogram per milliliter (h*ng/mL)
  R-PZO: number analyzed (Participants) | 17 | 9 | 9 | 2 | 14 | 15
  R-PZO | 1080 (1036) | 184 (150.0) | 2720 (1718) | NA (NA) — Mean and standard deviation was not calculated for participants fewer than 3 as per planned analysis. | 1190 (1110) | 907 (776.3)
  S-PZO: number analyzed (Participants) | 3 | 10 | 0 | 0 | 0 | 0
  S-PZO | 2.84 (0.9072) | 1240 (1124) |  |  |  |

ADVERSE EVENTS:
Time Frame: up to Day 40
Arm/Group | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/50 | 0/30 | 0/18 | 0/30 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/50 | 0/30 | 0/18 | 0/30 | 1/60
Other Adverse Events (participants affected / at risk) | 66/100 | 31/50 | 20/30 | 14/18 | 9/30 | 28/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg (N=100) | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg (N=50) | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg (N=30) | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg (N=18) | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg (N=30) | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg (N=60)
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1a: 4 to 6 Years L-PZQ ODT 50 mg/kg (N=100) | Cohort 1b: 4 to 6 Years Biltricide® 40 mg/kg (N=50) | Cohort 2: 2 to 3 Years L-PZQ ODT 50 mg/kg (N=30) | Cohort 3: 3 to 24 Months L-PZQ ODT 50 mg/kg (N=18) | Cohort 4a: 3 Months to 6 Years L-PZQ ODT 50 mg/kg (N=30) | Cohort 4b: 3 Months to 6 Years L-PZQ ODT 60 mg/kg (N=60)
Abdominal pain (Gastrointestinal disorders) | 23 | 10 | 9 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 18 | 3 | 4 | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 8 | 5 | 4 | 1 | 1 | 0
Somnolence (Nervous system disorders) | 8 | 3 | 8 | 2 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 8 | 4 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 1 | 1 | 3 | 0 | 3
Malaria (Infections and infestations) | 2 | 2 | 2 | 0 | 1 | 3
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 2
Rhinitis (Infections and infestations) | 5 | 0 | 0 | 0 | 1 | 0
Tinea capitis (Infections and infestations) | 3 | 3 | 2 | 1 | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 3 | 1 | 5 | 3
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 6 | 1 | 1 | 1 | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 5
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 0 | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Ketonuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3 | 1 | 4
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT03845140/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT03845140/SAP_001.pdf